CLINICAL TRIAL: NCT02667080
Title: Parameters of Sperm Quality in Consecutive Sperm Samples From Males Partners of Couples Seeking Treatment for Infertility
Brief Title: Sperm Quality in Consecutive Sperm Samples After 4-7 Days and 2 Hours of Sexual Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Hiva Alipour, Ph.D. Student, Research Assistant, Aalborg University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20140023
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Semen Quality
Keywords: Semen quality; Sexual Abstinence; sperm motility; DNA fragmentation
MeSH Terms: conditions — Sexual Abstinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ejaculate 1 (Active Comparator): Semen sample after 2-7 days of sexual abstinence
  Interventions: Other: 2-7 days of Sexual abstinence
- Ejaculate 2 (Active Comparator): Semen sample after 2 hours of sexual abstinence
  Interventions: Other: 2 hours of sexual abstinence

INTERVENTIONS:
Other: 2-7 days of Sexual abstinence — 2-7 days of Sexual abstinence
  Arms: Ejaculate 1
Other: 2 hours of sexual abstinence — 2 hours of sexual abstinence
  Arms: Ejaculate 2

SUMMARY:
The main purpose of the study is to assess to which degree a series of sperm parameters known to be associated with fertilization and implantation potential in artificial reproductive technology (ART) differ in consecutive sperm samples produced after 2-7 days and 2 hours of sexual abstinence in males from couples referring for ART treatment.

ELIGIBILITY:
Inclusion Criteria:

* male age between 18 and 50
* able to understand and read Danish

Exclusion Criteria:

* complete azospermia
* significant psychological illness
* significant cardiovascular disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Routine semen quality assessment | After liquefaction (30-35 minutes after ejaculation)
  Routine sperm quality check including Morphology, Motility and DNA fragmentation index using both the conventional manual method and computer assisted sperm analysis (CASA) systems.

SECONDARY OUTCOMES:
Outcome of ART treatments | up to one year after the sampling
  assessing and correlating the sperm quality with the results of the ART procedures

CONTACTS AND LOCATIONS:
Overall Officials: Ole Bjarane M.D., Ph.D., M.D., Ph.D., Study Director — Aalborg University Hospital, Gynecology Department; Hiva Alipour, D.V.M., Principal Investigator — Aalborg University, Faculty of Medicine, Department of Health Science and Technology; Fereshteh Dardmeh, D.V.M., Study Chair — Aalborg University, Faculty of Medicine, Department of Health Science and Technology; Gerhard Van DerHorst, Ph.D., Study Chair — University of the Western Cape, Capetown, South Africa; Christina Hnida, Ph.D., Study Chair — Aalborg University Hospital, Gynecology Department
Locations (1):
- Aalborg University Hospital, Dronninglund Fertility Clinic, Dronninglund, Denmark

IPD SHARING:
Plan to Share IPD: No